CLINICAL TRIAL: NCT04039204
Title: Elagolix for Fertility Enhancement Clinical Trial (EFFECT)
Brief Title: Elagolix for Fertility Enhancement Clinical Trial
Acronym: EFFECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00059474
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis; Unexplained Infertility
MeSH Terms: conditions — Endometriosis | interventions — elagolix; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elagolix (Experimental): Elagolix will be dosed at the higher dose used in pelvic pain trials, 200 mg twice a day for 2 months.
  Interventions: Drug: Elagolix
- Oral contraceptives (Ortho Cyclen) (Active Comparator): Elagolix will be compared to a less potent standard commonly used prior to IVF or embryo transfer, namely estrogen containing birth control pills.
  Interventions: Drug: Ortho Cyclen

INTERVENTIONS:
Drug: Elagolix — This orally active, reversible GnRH antagonist will be used to suppress endometriosis by lowering estrogen levels for 2 months prior to FET
  Other Names: Orilissa
  Arms: Elagolix
Drug: Ortho Cyclen — Oral contraceptive prescribed by physician.
  Arms: Oral contraceptives (Ortho Cyclen)

SUMMARY:
Studies suggest that undiagnosed endometriosis results in poor reproductive outcomes in the setting of In Vitro Fertilization and Embryo Transfer (IVF-ET). Biomarkers that predict endometriosis including B-cell lymphoma (BCL6) and Sirtuin 1 (SIRT1) are associated with reduced pregnancy rates following IVF-ET. Treatment with gonadotropin releasing hormone (GnRHr) receptor agonists (leuprolide acetate depot) has been shown to improve pregnancy rates following embryo transfer (ET). In this randomized controlled trial, a new generation GnRHr antagonist, elagolix, will be compared to oral contraceptives (OCPs) for suppression of suspected endometriosis prior to ET. Both groups will receive two months of treatment prior to frozen embryo transfer of a single euploid embryo. Outcomes will include pregnancy rate, miscarriage rate and ongoing and live birth rate following treatment. Patients experiencing unanticipated problems or who experience adverse events such that they do not tolerate the treatment they are assigned, will be allowed to discontinue treatment and be provided the opportunity to use the other treatment if they so choose. The outcomes of such cycles would be collected separately and included as observational data only and not included in the randomized data analysis. Alternatively, they can simply drop out of the study and resume medical therapy as appropriate or pursue frozen embryo transfer as previously planned.

DETAILED DESCRIPTION:
Although meta-analyses have not demonstrated an effect of endometriosis on IVF outcomes, most women with endometriosis undergoing IVF have not been diagnosed or treated for their disease. Recent evidence suggests that biomarkers for endometriosis predict IVF failure and miscarriage. Further suppression of endometriosis prior to IVF has been shown to dramatically improve pregnancy rates in unexplained infertility with suspected endometriosis. Elagolix (Orilissa) is a new generation FDA approved orally active GnRHr antagonist that is rapidly reversible, for the treatment of endometriosis and pelvic pain. There have been no studies on the efficacy of elagolix for the treatment of endometriosis-associated infertility. Given the recent study in Fertility and Sterility demonstrating IVF outcome prediction using BCL6 as a biomarker for the presence of endometriosis and subsequent preliminary data showing benefit using surgery and GnRH agonist therapy, there is adequate rationale to examine the use of the orally active, non-peptide compound (elagolix) for estrogen suppression prior to frozen embryo transfer in women who test positive for BCL6 and an associated protein, SIRT1. In this multi-central randomized controlled trial (RCT), the EFFECT Trial, the investigators plan to recruit 100 subjects with prior unexplained IVF failure with positive endometrial BCL6/SIRT1 expression. To qualify all subjects will need to have a preimplantation genetic testing (PGT-A) tested euploid embryo and intentions to undergo frozen embryo transfer. Subjects will be randomized to receive elagolix (200 mg BID) or OCPs for 2 months prior to standardized FET. Primary study outcomes will be pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Anti-Mullerian Hormone (AMH) > 0.5 and < 10
* At least 1 euploid embryo for transfer
* Prior endometrial biopsy showing elevated BCL6 and SIRT1 expression
* Endometrial thickness > 5.9 and < 14 mm

Exclusion Criteria:

* Uterine fibroids > 4 cm (intramural)
* Polycystic ovary syndrome (Rotterdam criteria)
* Ovarian failure and donor eggs or oocytes
* Positive lupus anticoagulant or positive anti-cardiolipin antibody testing
* Diabetes mellitus (Type I or II)
* Untreated hypothyroidism
* Untreated hyperprolactinemia
* BMI <17 or > 35
* Uncorrected uterine anomaly

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women with infertility seeking embryo transfer are eligible to participate
Enrollment: 10 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Lessey, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Univesity Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor HS, Giudice LC, Lessey BA, Abrao MS, Kotarski J, Archer DF, Diamond MP, Surrey E, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Rowan JP, Duan WR, Ng J, Schwefel B, Thomas JW, Jain RI, Chwalisz K. Treatment of Endometriosis-Associated Pain with Elagolix, an Oral GnRH Antagonist. N Engl J Med. 2017 Jul 6;377(1):28-40. doi: 10.1056/NEJMoa1700089. Epub 2017 May 19. PMID 28525302
- [Background] Surrey E, Taylor HS, Giudice L, Lessey BA, Abrao MS, Archer DF, Diamond MP, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Singh SS, Rechberger T, Agarwal SK, Duan WR, Schwefel B, Thomas JW, Peloso PM, Ng J, Soliman AM, Chwalisz K. Long-Term Outcomes of Elagolix in Women With Endometriosis: Results From Two Extension Studies. Obstet Gynecol. 2018 Jul;132(1):147-160. doi: 10.1097/AOG.0000000000002675. PMID 29889764
- [Background] Likes CE, Cooper LJ, Efird J, Forstein DA, Miller PB, Savaris R, Lessey BA. Medical or surgical treatment before embryo transfer improves outcomes in women with abnormal endometrial BCL6 expression. J Assist Reprod Genet. 2019 Mar;36(3):483-490. doi: 10.1007/s10815-018-1388-x. Epub 2019 Jan 4. PMID 30610661
- [Background] Almquist LD, Likes CE, Stone B, Brown KR, Savaris R, Forstein DA, Miller PB, Lessey BA. Endometrial BCL6 testing for the prediction of in vitro fertilization outcomes: a cohort study. Fertil Steril. 2017 Dec;108(6):1063-1069. doi: 10.1016/j.fertnstert.2017.09.017. Epub 2017 Nov 7. PMID 29126613
- [Background] Littman E, Giudice L, Lathi R, Berker B, Milki A, Nezhat C. Role of laparoscopic treatment of endometriosis in patients with failed in vitro fertilization cycles. Fertil Steril. 2005 Dec;84(6):1574-8. doi: 10.1016/j.fertnstert.2005.02.059. PMID 16359945

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elagolix | Oral Contraceptives (Ortho Cyclen)
Started | 5 | 5
Completed | 5 | 3
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elagolix | Oral Contraceptives (Ortho Cyclen) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9699175 (3.894399758) | 32.417758 (3.606106781) | 34.44094 (4.236217486)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Live Births
Time Frame: Month 9
Measure: Number; unit: live births
Arm/Group | Elagolix | Oral Contraceptives (Ortho Cyclen)
Number analyzed (Participants) | 5 | 3
live births | 3 | 1

2. Secondary Outcome: Number of Miscarriages
Description: The number of subjects with a first trimester pregnancy loss
Time Frame: week 15
Population: Out of three participants who had embryo transfers in Ortho Cyclen arm, two had viable pregnancies. One of those two had a live birth and one of those two had a miscarriage. So only two participants were analyzed in the Ortho Cyclen arm for this outcome.
Measure: Number; unit: miscarriages
Arm/Group | Elagolix | Oral Contraceptives (Ortho Cyclen)
Number analyzed (Participants) | 5 | 2
miscarriages | 2 | 1

3. Secondary Outcome: Number of Viable Pregnancies
Time Frame: 12 to 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Elagolix | Oral Contraceptives (Ortho Cyclen)
Number analyzed (Participants) | 5 | 3
Participants | 5 | 2

4. Other Pre Specified Outcome: Inflammation Measurements
Description: nanostring arrays for both miRNAs and inflammation biomarkers
Time Frame: week 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: baseline through month 9
Arm/Group | Elagolix | Oral Contraceptives (Ortho Cyclen)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elagolix (N=5) | Oral Contraceptives (Ortho Cyclen) (N=5)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04039204/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT04039204/ICF_000.pdf